CLINICAL TRIAL: NCT04866368
Title: Comparison of Sacral Erector Spinae Plane Block and Dorsal Penile Block in Pain Management in Patients Undergoing Hypospadias Surgery
Brief Title: Comparison of Erector Spinae Plane Block and Penile Block in Hypospadias Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Can AKSU, Associate professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KSU 2019/12-17
Record Dates: First submitted 2021-04-27; First posted 2021-04-29 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Postoperative Pain; Analgesia
Keywords: Regional anaesthesia; Pediatric anesthesia; Erector spinae plane block; Penil block
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The erector spinae plane block (Active Comparator): The ultrasound-guided Erector spinae plane block (ESPB) with 1 ml/kg 0,25 % bupivacaine at the lumbar vertebral level will perform before surgery to all patients in the ESPB group.
  Interventions: Procedure: The ultrasound-guided Sacral Erector spinae plane block
- The penile block (Active Comparator): The penile block with 0,5ml/kg 0,25 % bupivacaine will be performed after the patients give standard general anesthesia and a laryngeal mask is applied.
  Interventions: Procedure: The dorsal penile block

INTERVENTIONS:
Procedure: The ultrasound-guided Sacral Erector spinae plane block — postoperative pain procedure
  Arms: The erector spinae plane block
Procedure: The dorsal penile block — postoperative pain procedure
  Arms: The penile block

SUMMARY:
In this study, we aimed to compare ultrasound-guided sacral erector spinae plane block and dorsal penile block on postoperative analgesic effect in hypospadias surgery.

DETAILED DESCRIPTION:
ASAI-II, 1-9 years old patients with hypospadias diagnosis and operated in Kahramanmaraş Sütçü İmam University hospital and Kocaeli University hospital were randomized with closed envelope technique and divided into two groups as penile block or erector spinae plane block. Erector spinae plane block or penile block application (by Gözen Öksüz, Can Aksu) will be performed after the patients give standard general anesthesia and a laryngeal mask is applied. Vital signs such as pulse, sp02, blood pressure will be monitored before, during and at the end of the operation. At the end of the operation and after the patient is awakened 5. min., 30 min. 1., 2., 4., 6., 12., 24. hourly FLACC pain scores, number of analgesic use within 24 hours, patient family satisfaction (1: dissatisfied, 2: satisfied, 3: very satisfied), complication rates will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology Classification (ASA) I-II, 1-9 years aged patients patients who scheuled elective hypospadias surgery in Kahramanmaraş Sütçü İmam University Hospital and Kocaeli University Hospital

Exclusion Criteria:

* American Society of Anesthesiology Classification (ASA) III-IV, patients with coagulopathy patients with infection at the injection site

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-04-20 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
FLACC score | during postoperative 24 hour
  At the end of the operation and after the patient is awakened 5th min., 30th min., 1st, 2nd, 4th, 6th, 12th, 24th Hourly FLACC pain scores will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Kocaeli University Hospital, İzmit, Kocaeli
  - Kahramanmaras Sütcü Imam University, Kahramanmaraş

REFERENCES:
- See also: Sacral Erector Spinae Plane Block with longitudinal midline approach: Could it be the new era for pediatric postoperative analgesia? — https://pubmed.ncbi.nlm.nih.gov/31203111/